CLINICAL TRIAL: NCT00103103
Title: A Phase II Combination Trial of PS-341 and 5-FU/LV in Gastric and/or GE Junction Adenocarcinoma
Brief Title: Bortezomib, Fluorouracil, and Leucovorin in Treating Patients With Metastatic or Unresectable Stomach Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000410827; CCC-PHII-43; NCI-5991; LAC-USC-3G036
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Bortezomib; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: bortezomib
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with fluorouracil and leucovorin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with fluorouracil and leucovorin works in treating patients with metastatic or unresectable stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine response in patients with previously treated metastatic or unresectable gastric or gastroesophageal junction adenocarcinoma treated with bortezomib, fluorouracil, and leucovorin calcium.

Secondary

* Determine time to progression and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 8, and 15. One hour after completion of bortezomib, patients receive leucovorin calcium IV and fluorouracil IV followed by fluorouracil IV continuously over 46 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for survival.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gastric or gastroesophageal junction adenocarcinoma

  * Metastatic or unresectable disease
* Progressive disease after receiving 1 prior chemotherapy regimen for metastatic disease comprising 1 of the following:

  * Fluorouracil
  * Cisplatin and irinotecan
  * Capecitabine
  * Taxanes
* Measurable disease
* No esophageal cancer
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No acute ischemia by EKG
* No significant conduction abnormality by EKG, including either of the following:

  * Bifasicular block, defined as left anterior hemiblock in the presence of right bundle branch block
  * Second or third degree atrioventricular block
* No history of cardiac or cerebrovascular disease due to hypotension and tachycardia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 6 months after study participation
* No ongoing or active infection
* No other uncontrolled illness
* No peripheral neuropathy ≥ grade 2 within the past 2 weeks
* No allergy to boron or mannitol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* More than 2 weeks since prior major surgery

Other

* No concurrent highly active anti-retroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST every 8 weeks

SECONDARY OUTCOMES:
Time to progression every 8 weeks
Overall survival
Toxicity every 4 weeks
Molecular correlates on and off study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania